CLINICAL TRIAL: NCT03286985
Title: The Prevalence and Incidence of Deep Venous Thrombosis in General ICU Patients Receiving Enoxaparine Prophylaxis
Brief Title: The Prevalence and Incidence of DVT in General ICU
Acronym: preTIME
Status: Completed | Type: Observational
Sponsor: Masaryk Hospital Krajská zdravotní a.s. (Other)
Responsible Party: Principal Investigator, Jan Benes, MUDr. Ing., Masaryk Hospital Krajská zdravotní a.s.
Other Study IDs: 236/60
Record Dates: First submitted 2016-05-10; First posted 2017-09-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-03

CONDITIONS: Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General ICU patients: No intervention is associated with inclusion to the study (observational study). Included will be all patients admitted to general ICU with ICU stay >72 hours, having deep venous thrombosis prophylaxis appropriate to clinical setting and following the recent guidelines. All study participants will undergo repeated noninvasive ultrasound testing for deep venous thrombosis, which is normal part of the routine care in our ICU.

SUMMARY:
Deep venous thrombosis (DVT) represents a major problem in intensive care unit (ICU) patients. Despite the use of recommended pharmacological prophylaxis with low molecular weight heparin (LMWH), the incidence of DVT during ICU stay has been reported between 5 and 15 %. The incidence may vary due to many factors, for example the type of ICU population, the type of protocol of pharmacological prophylaxis and also the type of diagnostic approach. Before formerly planned clinical study targeted to lower DVT incidence by individualizing the dose of LMWH, the investigators decided to evaluate the real DVT incidence in the investigated ICU. The prevalence and incidence will be assessed by ultrasound testing in general ICU patients. on the sample of 200 patients. The investigators hypothesize DVT incidence of 5 %. The compliance to the local DVT prophylaxis protocol will be also evaluated.

DETAILED DESCRIPTION:
Type of the study: Observational prospective cohort study. Hypothesis: Despite appropriate prophylaxis of deep venous thrombosis in general ICU patients in accordance with the current guidelines, the incidence of deep venous thrombosis is 5 - 10%.

Sample size: 200 consecutive general ICU patients. Inclusion and exclusion criteria: defined in the Eligibility section. Protocol description: All patients admitted to ICU with expected period of the stay longer than 72 hours will be evaluated for the presence of deep venous thrombosis by ultrasound testing during the first 48 hours of ICU stay. Thereafter, each participant will be examined by ultrasound testing twice a week until the discharge from ICU. All patients will receive deep venous thrombosis prophylaxis following the current guidelines. All patients with positive finding of deep venous thrombosis will be managed in accordance with the current guidelines.

Ultrasound examination for deep venous thrombosis: Ultrasound compression test at the following locations: common femoral vein at the groin, deep femoral vein, popliteal vein, both extremities.

ELIGIBILITY:
All general ICU patients meeting exclusion and inclusion criteria.

Inclusion criteria:

1. General ICU patient with expected length of stay more than 72 hours

Exclusion Criteria:

1. Inability to perform ultrasound investigation for deep venous thrombosis (for medical or technical reasons)
2. ICU stay shorter than 72 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of deep venous thrombosis | 24 hours from ICU admission to ICU discharge (up to 12 month)
  Number of patients with new onset deep venous thrombosis diagnosed during ICU stay (ie deep venoous thrombosis developed after the first 24 hours of ICU stay)

SECONDARY OUTCOMES:
Prevalence of deep venous thrombosis | From ICU admission to ICU discharge (up to 12 month)
  A number of patients with deep venous thrombosis diagnosed anytime during ICU stay (on admission and during ICU stay)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Beneš, MD, Principal Investigator — Department of Anesthesiology, Perioperative Medicine and Intensive Care, J.E. Purkinje University, Masaryk Hospital in Usti nad Labem, Usti nad Labem, Czech Republic
Locations (1):
- Masaryk Hospital, Ústí nad Labem, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Qaseem A, Chou R, Humphrey LL, Starkey M, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Venous thromboembolism prophylaxis in hospitalized patients: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2011 Nov 1;155(9):625-32. doi: 10.7326/0003-4819-155-9-201111010-00011. PMID 22041951
- [Derived] Benes J, Skulec R, Jobanek J, Cerny V. Fixed-dose enoxaparin provides efficient DVT prophylaxis in mixed ICU patients despite low anti-Xa levels: A prospective observational cohort study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2022 May;166(2):204-210. doi: 10.5507/bp.2021.031. Epub 2021 May 27. PMID 34042098